CLINICAL TRIAL: NCT00180752
Title: The Investigation of HDAC and NF Kappa B Activity in Peripheral Skeletal Muscle in COPD
Brief Title: HDAC Activity in Peripheral Skeletal Muscle in COPD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Michael Polkey, Professor of Respiratory Medicine, Imperial College London
Other Study IDs: MusHDAC -1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2008-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma and serum samples, quadriceps muscle specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
We wish to study the effect of Chronic Obstructive Pulmonary Disease on the activity of the nuclear transcription pathway in peripheral skeletal muscle to determine whether altered activity of this pathway may be responsible for the muscle dysfunction observed in these patients.

DETAILED DESCRIPTION:
Peripheral muscle dysfunction is well recognised in COPD. We wish to study patients who we have found to have weak quadriceps muscles and study the molecular mechanisms underlying this problem. Patients will be well characterised with regard to their physiologic parameters and quadriceps muscle biopsies will be taken. These biopsy samples will be analysed with respect to NFkappaB activity and HDAC activity by nuclear extraction and for muscle inflammatory cytokines. We know that in the lung tissue of COPD patients there is evidence of a reduction in HDAC activity which might be responsible for the higher levels of pronflammatory cytokines in the lung. We will also study a healthy control group and a small selection of patients who are in respiratory failure due to idiopathic scoliosis in the same way.

ELIGIBILITY:
Inclusion Criteria:

COPD

-

Exclusion Criteria:

Aspirin therapy Bleeding diasthesis Neuromuscular disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients and healthy age-and sex-matched controls
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Polkey, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agusti A, Morla M, Sauleda J, Saus C, Busquets X. NF-kappaB activation and iNOS upregulation in skeletal muscle of patients with COPD and low body weight. Thorax. 2004 Jun;59(6):483-7. doi: 10.1136/thx.2003.017640. PMID 15170030
- [Background] Ito K, Ito M, Elliott WM, Cosio B, Caramori G, Kon OM, Barczyk A, Hayashi S, Adcock IM, Hogg JC, Barnes PJ. Decreased histone deacetylase activity in chronic obstructive pulmonary disease. N Engl J Med. 2005 May 12;352(19):1967-76. doi: 10.1056/NEJMoa041892. PMID 15888697